CLINICAL TRIAL: NCT05846919
Title: High Flow Oxygen in Preoxygenation During Rapid Sequence Induction in Infants and Small Children: Pilot Randomized Controlled Trial
Brief Title: High Flow Oxygen in Preoxygenation During Rapid Sequence Induction in Infants and Small Children
Acronym: PRSIHFO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KDAR PRSI-START-UP
Record Dates: First submitted 2023-04-17; First posted 2023-05-06 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Rapid Sequence Induction (RSI); Preoxygenation
Keywords: Rapid sequence induction (RSI); High flow nasal oxygenation (HFNO); High flow nasal cannula (HFNC); preoxygenation; children; pediatric; infant

STUDY DESIGN:
Intervention Model Description: Triple group randomized controlled pilot trial
Who Masked: Participant
Masking Description: Participant under general anesthesia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pediatric patients indicated for RSI and face-mask preoxygenation (Active Comparator): face-mask preoxygenation (flow 2 L/kg/minute, max 6 L/minute) with 100 % oxygen for three minutes.
  Interventions: Procedure: face-mask preoxygenation
- Pediatric patients indicated for RSI and HFNOC preoxygenation (Active Comparator): HFNOC preoxygenation (flow 2 L/kg/minute, max 6 L/minute) with 100 % oxygen for three minutes.
  Interventions: Procedure: HFNOC preoxygenation
- Pediatric patients indicated for RSI and HFNOC + face-mask preoxygenation (Experimental): HFNOC (flow 2 L/kg/minute) + face-mask preoxygenation (flow 2 L/kg/minute, max 6 L/minute) - with 100 % oxygen for three minutes.
  Interventions: Procedure: HFNOC + face-mask preoxygenation

INTERVENTIONS:
Procedure: face-mask preoxygenation — face-mask preoxygenation (flow 2 L/kg/minute, max 6 L/minute) with 100 % oxygen for three minutes.
  Arms: Pediatric patients indicated for RSI and face-mask preoxygenation
Procedure: HFNOC preoxygenation — HFNOC preoxygenation (flow 2 L/kg/minute, max 6 L/minute) with 100 % oxygen for three minutes.
  Arms: Pediatric patients indicated for RSI and HFNOC preoxygenation
Procedure: HFNOC + face-mask preoxygenation — HFNOC (flow 2 L/kg/minute) + face-mask preoxygenation (flow 2 L/kg/minute, max 6 L/minute) - with 100 % oxygen for three minutes.
  Arms: Pediatric patients indicated for RSI and HFNOC + face-mask preoxygenation

SUMMARY:
Airway management is crucial part of the anaesthesia. There is always a considerable risk of complications or even failure during the anaesthesia induction and airway management. The risk could be greater considering anaesthesia in children and neonates because of their anatomical and physiological differences. Children and neonates are more susceptible to hypoxia and bradycardia during induction of anaesthesia, this risk is even greater during the rapid sequence induction/intubation (RSI), in which there is an apnoeic pause because of the absence of manual ventilation. Because of the pause it is necessary to provide enough oxygen in advance during preoxygenation. The aim of this trial is to compare providing oxygen by face-mask and by high-flow nasal oxygen cannula. Another outcome is to evalute the safety profile RSI in children and neonates.

DETAILED DESCRIPTION:
All patients requiring an acute surgery and rapid sequence induction/intubation will be checked for eligibility criteria and then an informed consent will be obtained. Afterwards, randomization will take place, which will divide a patient into one of three groups: 1) RSI + face-mask preoxygenation, 2) RSI + high-flow nasal oxygen cannula (HFNOC) preoxygenation and 3) RSI + face-mask and HFNOC preoxygenation.

The demographic data, type of surgery and vital signs will be observed. Primary outcomes will be the impact of HFNOC preoxygenation on oxygen saturation by pulse oximetry (SpO2) and heart rate during the induction of anaesthesia. Secondary outcomes will be safety of the RSI protocol, Cormack-Lehane score, incidence of difficult airway management, number of the intubation attempts and episodes of regurgitation/aspiration.

RSI will be done according to our protocol. Initially, equipment will be checked and an i.v. line will be checked/started and then a bolus of ketamine will be given (0,2-0,5 mg/kg intravenously,) for the face-mask/HFNOC tolerance and the table will be tilted to anti-Trendelenburg position. In case of difficult or unable of intravenous line insertion, intramuscular bolus of ketamin (1-3mg/kg i.m.) could be used prior to another attempt. Afterward, the preoxygenation will start according to the randomization result - group 1) face-mask preoxygenation (flow 2 L/kg/minute, max 6 L/minute), group 2) HFNOC preoxygenation (flow 2 L/kg/minute, max 6 L/minute) and group 3) HFNOC (flow 2 L/kg/minute) + face-mask preoxygenation (flow 2 L/kg/minute, max 6 L/minute) - with 100 % oxygen for three minutes. Then a bolus of anaesthetic and myorelaxant agent will be given (propofol 2,5 mg/kg in haemodynamically stable, ketamine in haemodynamically unstable and rocuronium 1 mg/kg or suxamethonium 1,5 mg/kg if sugammadex bolus was given in last 24 hours). The neuromuscular blockade will be monitored, first intubation attempt will start as soon as single twitch will be bellow 10 % or train-of-four (TOF) bellow 1 or after 60 seconds, whichever comes first. After that, the first intubation attempt will take place, a video laryngoscopy will be used and Cormack-Lehane score will be documented photographically. The attempt will end either by successful intubation with monitored capnography wave or by failure.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients indicated for rapid sequence induction
* informed consent

Exclusion Criteria:

* decline to participate
* rapid sequence induction not required for anesthesia induction

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of desaturation under 90% | Intraoperatively
  peripheral oxygen saturation measured by saturation probe will be evaluated and the saturation at the moment of first successful intubation attempt (defined by the first capnography tracing), the incidence of saturation declined below 90% will be recorded
Incidence of manual ventilation during RSI | Intraoperatively
  incidence of manual ventilation during preoxygenation due to desaturation will be evaluated

SECONDARY OUTCOMES:
Incidence of desaturation under 80% | Intraoperatively
  peripheral oxygen saturation measured by saturation probe will be evaluated and the saturation at the moment of first successful intubation attempt (defined by the first capnography tracing), the incidence of saturation declined below 90% will be recorded
time to desaturation under 90% | Intraoperatively
  peripheral oxygen saturation measured by saturation probe will be evaluated and the saturation at the moment of first successful intubation attempt (defined by the first capnography tracing), the time to reach saturation below 90% will be recorded
time to desaturation under 80% | Intraoperatively
  peripheral oxygen saturation measured by saturation probe will be evaluated and the saturation at the moment of first successful intubation attempt (defined by the first capnography tracing), the time to reach saturation below 80% will be recorded
time needed for relaxation | Intraoperatively
  time between the induction dose and the optimal intubation conditions (defined by accelerometry - single twitch below 10%, or TOF below 1, or post-tetanic count - PTC tracing) will be recorded
time needed for intubation | Intraoperatively
  time between the induction dose and first capnography tracing will be recorded
time to reach oxygen saturation 100% | Intraoperatively
  time between the preoxygenation initiation and the 100% oxygen saturation between the groups will be recorded
First intubation attempt success rate | Intraoperatively
  First intubation attempt success rate
Number of intubation attempts to successful intubation | Intraoperatively
  Number of intubation attempts to successful intubation
Intubation conditions | Intraoperatively
  Intubation conditions defined by Cormack-Lehane score
Incidence of complications | Intraoperatively
  Incidence of complications - aspiration, regurgitation, difficult intubation

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided